CLINICAL TRIAL: NCT01833715
Title: Efficacy Methadone for Management Postoperative Pain After the Use of Anesthesia Intravenous in Laparoscopic Cholecystectomy
Brief Title: Methadone for Postoperative Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Valparaiso (Other)
Responsible Party: Principal Investigator, Eva Madrid, Investigator, Universidad de Valparaiso
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P03/13
Record Dates: First submitted 2013-03-30; First posted 2013-04-17 (Estimated); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Pain, Postoperative
Keywords: Pain, Postoperative; Analgesics, Opioid; Methadone; Morphine
MeSH Terms: conditions — Pain, Postoperative | interventions — Morphine; Methadone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Morphine (Active Comparator): morphine group 0.08 mg / kg, to start surgery
  Interventions: Drug: Morphine; Drug: TIVA
- Methadone (Experimental): methadone group 0.08 mg / kg, to start surgery
  Interventions: Drug: Methadone; Drug: TIVA

INTERVENTIONS:
Drug: Morphine — Morphine group,receive morphine 0.08 mg / kg at the start of surgery
  Arms: Morphine
Drug: Methadone — Methadone group,receive methadone 0.08 mg / kg at the start of surgery
  Arms: Methadone
Drug: TIVA — TIVA: General anesthesia will be based on Remifentanil and Propofol (TIVA-TCI), titrated to achieve bispectral index (BIS) between 40 and 60.

SUMMARY:
The aim of this study is to compare the efficacy of methadone versus morphine in dealing with postoperative pain, in laparoscopic cholecystectomy under total intravenous anesthesia (TIVA); Efficacy is defined in terms of the difference of milligrams in morphine used as rescue analgesia postoperatively. Our hypothesis is that methadone is more effective than morphine for postoperative pain treatment.

DETAILED DESCRIPTION:
Patients undergo laparoscopic cholecystectomy at Almirante Nef Naval Hospital will be recruited, between March and July 2013. The sample size was calculated to obtain an average difference of 4 mg of morphine (DE 1.5) to 3 mg of morphine (DE 1.5), with a power of 80% and a significance level of 0.05. This came down to 36 randomized patients into each group, so 86 patients will be recruited considering a 15% loss to follow up.

Before signing an informed consent, we will explain to them how to classify pain intensity numerical rating scale (NRS) and this will be evaluated periodically during the first 24 hours after surgery.

General anesthesia will be based on Remifentanil and Propofol, titrated to achieve bispectral index (BIS) between 40 and 60. Patients will be randomized into methadone group (ME) and morphine group (MO), they will receive 0.08 mg / kg bolus of methadone or 0.08 mg / kg bolus of morphine as applicable at the time of beginning surgery. Postoperative analgesia will be standard for both groups. Patient´s demographic data will be filed as well as surgical timings.

All patients will remain in the anesthetic recovery room for the first two hours , to get a record taken of vital signs and measurement of NRS at 5, 15, 30, 60 and 120 minutes. If NRS is greater than or equal to 4, 1 mg of morphine ev will be used as analgesic rescue. In room measuring NRS continue hospitalized at 4, 8, 12 and 24 hours postoperatively and were used as rescue analgesia if ketorolac 30mg ev NRS is greater than or equal to 4. The amount of morphine is registered and ketorolac rescue of both groups as well as pain assessment scores. The occurrence of adverse effects such as nausea, vomiting, pruritus, urinary retention and respiratory depression is also recorded in both groups, to be compared later as a secondary objective.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing laparoscopic cholecystectomy in the Almirante Nef Naval Hospital
* Patients ASA 1 or 2

Exclusion Criteria:

* Patients with renal insufficiency (creatinine> 2.0 mg / dl)
* Patients with a history of liver failure
* Patients with BMI> 35 kg/m2
* Patients with hypersensitivity to the drugs in question
* History of chronic use of opioids
* Need for conversion to open surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Difference in milligrams of morphine used as rescue analgesia | First 24 hours postoperatively
  Difference in milligrams of morphine used as rescue analgesia in postoperative period in both groups

SECONDARY OUTCOMES:
Difference in pain scores, using the Numeric Rating Scale | First 24 hours postoperatively
  Difference in pain scores, using the Numeric Rating Scale at 5, 15, 30, 60 and 120 minutes postoperative. Also at 4, 8, 12 and 24 hours postoperatively, during hospitalization.

OTHER OUTCOMES:
The different of the adverse effect | First 24 hours postoperatively
  The total number of adverse effects such as nausea, vomiting, pruritus, urinary retention and respiratory depression is recorded in both groups, to be compared later as a secondary objective.

CONTACTS AND LOCATIONS:
Overall Officials: NICOLAS ARRIAZA, Physician, Principal Investigator — University Valparaiso
Locations (1):
- Almirante Nef Naval Hospital, Viña del Mar, Región de Valparaíso, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arriaza N, Papuzinski C, Kirmayr M, Matta M, Aranda F, Stojanova J, Madrid E. Efficacy of methadone for the management of postoperative pain in laparoscopic cholecystectomy: A randomized clinical trial. Medwave. 2021 Mar 23;21(2):e8135. doi: 10.5867/medwave.2021.02.8134. English, Spanish. PMID 33905405